CLINICAL TRIAL: NCT03687411
Title: Development of an Ultrasound Guided Automated Spinal Landmark Identification System (uSINE Study)
Brief Title: An Ultrasound Guided Automated Spinal Landmark Identification System
Acronym: uSINE
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: KK Women's and Children's Hospital (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: NHIC-I2D-1708180
Record Dates: First submitted 2018-08-22; First posted 2018-09-27 (Actual); Last update posted 2024-10-09 (Actual); Status verified 2024-10

CONDITIONS: Spinal Anaesthesia; Obesity
Keywords: spinal anaesthesia; Neuraxial ultrasonography; landmark identification
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- ULTRA-SINE (phases 1-4) (Experimental): There will be four phases in this proposed uSINE system. In first phase attending anaesthetist will use the automated spinal landmark system for neuraxial needle insertion to place the neuraxial anaesthesia in non-obese patients.
  For the second phase, obese patients will have ultrasound scan of their lumbar back and no needle insertion is involved.
  In third phase, conventional ultrasonography is used prior to the needle insertion, and needle insertion is conducted manually as per routine practice. The images collected in the system will be used for annotation and evaluation which serves as training material for uSINE to optimize its algorithm to improve landmark identification for obese patients. The fourth phase will have uSINE system used prior to the needle insertion, with the neuraxial needle insertion conducted manually as per routine practice. The identification accuracy and first-attempt puncture success rate of uSINE will be determined.
  Interventions: Procedure: Neuraxial ultrasonography

INTERVENTIONS:
Procedure: Neuraxial ultrasonography — Ultrasound gel is applied to lower back lumbar spine of patient and placed with an ultrasound probe around the sacral region. The graphical interface of the software integrated with ultrasound machine will help identify the sacrum. The probe is moved in until the L3/4 interspinous space is identified for skin surface marking. Once the longitudinal scan is completed, the investigator will turn the probe 90° clockwise for transverse scan to identify ligamentum flavum.

SUMMARY:
Neuraxial ultrasonography has been shown a safe and effective technique to enhance the overall success rate of lumbar puncture and reduce the number of injection attempts. However, the current blind palpation landmark technique is known to be highly inaccurate and may increase the risk of multiple insertion attempts, patient suffering and complication rates such as spinal cord injury. Various clinical studies have confirmed the effectiveness of ultrasound imaging compared with the traditional palpation method. However, none of the present system can achieve real-time guidance.

The overall aim of this proposal is to develop an ultrasound guided automated spinal landmark identification with real-time neuraxial needle insertion system (uSINE) to improve patient safety and efficacy of neuraxial procedure needle insertion success. This will be achieved in 4 phases of technology development and clinical trial phases. The investigators will recruit 20 subjects in a prospective cohort study to investigate the spinal needle first attempt success rate as a clinically relevant outcome. The secondary aim is to develop an automated spinal landmark identification algorithm using image processing to identify spinal landmarks in 50 obese patients. Third phase objective will be to obtain clinical data, and evaluation and annotation of the clinical data of spinal ultrasonography in 65 obese patients (BMI > 30kg/m2), whereas the fourth phase will measure the uSINE identification accuracy and first-attempt puncture success rate of uSINE in a clinical study of 65 obese patients (BMI > 30kg/m2).

DETAILED DESCRIPTION:
This is a prospective cohort study to evaluate the efficacy and accuracy of ultrasound guided automated spinal landmark identification with real-time neuraxial needle insertion system (uSINE).

The subjects assume a seated position and the lower back is exposed. Ultrasound gel will be applied to the lower back lumbar spine and the investigator will place an ultrasound curved array probe around the sacral region. The graphical interface of the software, integrated with the wireless ultrasound probe and ultrasound machine, will inform the investigator when the software has positively identified the sacrum. The investigator will then move the probe in a steady vertical upward longitudinal direction until the L3/4 interspinous space is identified by the program. The ultrasound algorithm will identify the skin surface marking. The longitudinal section of the scan will be completed and the investigator will turn the probe 90 degrees clockwise around the probe center to the transverse view.

The transverse scan consists of minimal vertical movements by the investigator who will obtain images using the ultrasound probe. The software will signal when the correct identification of the ligamentum flavum is visualized. The scan sequence will be completed.

The first phase will involve 20 non-obese patients who are undergoing neuraxial anaesthesia or analgesia. The system is used prior and during needle insertion to provide real-time guidance for the anaesthetists. The neuraxial needle insertion is conducted manually by the anaesthetist as per routine practice.

In the second phase, 50 obese patients (body mass index more than 30) will be recruited to investigate and develop an "obesity" mode visualisation of the ultrasound guided automated spinal landmark identification. This will be to advance the technology to evaluate more difficult anatomy and more complex neuraxial needle insertion in future work plan. The patients' back will be scanned to obtain the images. The neuraxial needle insertion is conducted manually (i.e. independent of the ultrasound results) by the anaesthetist as per hospital routine practice.

The third phase involve data collection and annotation of spinal ultrasonography in 65 obese patients, followed by a fourth phase to measure the uSINE identification accuracy and first-attempt puncture success rate in 65 obese patients.

ELIGIBILITY:
Inclusion Criteria:

First phase:

* Age 21 - 75 years old patients who require neuraxial anesthesia for surgical procedure;
* Normal body mass index (Weight 40-90 kg, Height 140-180cm).

Second-fourth phases:

* Obese patients aged between 21-75 years old;
* body mass index more than 30.

Exclusion Criteria:

* History of scoliosis;
* History of spinal instrumentation;
* Drug allergy to ultrasound transmission gel;
* Visible wound or injury in the lumbar spine.

Ages: 21 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Only female undergoing surgery in the institution will be recruited (the mentioned institution provides healthcare services only to women and children)
Enrollment: 200 (Estimated)
Dates: Start 2018-05-24 (Actual); Primary Completion 2026-10-14 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
First attempt success rate of spinal anaesthesia | 12 hours
  The rate of cases achieving successful spinal anaesthesia at first attempt of insertion

SECONDARY OUTCOMES:
Number of spinal attempts | 12 hours
  The number of attempts to achieve successful spinal anaesthesia
Time taken for ligamentum flavum identification | 12 hours
  Time taken to identify the ligamentum flavum in the transverse view
Distance from skin to ligamentum flavum | 12 hours
  Distance from skin to ligamentum flavum as detected by the algorithm

CONTACTS AND LOCATIONS:
Overall Officials: Ban L Sng, FANZCA, Principal Investigator — KK Women's and Children's Hospital
Locations (1):
- KK Women's and Children's Hospital, Singapore, Singapore

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] In Chan JJ, Ma J, Leng Y, Tan KK, Tan CW, Sultana R, Sia ATH, Sng BL. Machine learning approach to needle insertion site identification for spinal anesthesia in obese patients. BMC Anesthesiol. 2021 Oct 18;21(1):246. doi: 10.1186/s12871-021-01466-8. PMID 34663224

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-08-08): https://cdn.clinicaltrials.gov/large-docs/11/NCT03687411/Prot_SAP_001.pdf